CLINICAL TRIAL: NCT04482296
Title: Effect of Zinc Supplementation on Depression in Selective Serotonin Reuptake Inhibitors-treated Major Depressive Disorder Patients
Brief Title: Effect of Zinc Supplementation on Depression in SSRI-treated Major Depressive Disorder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Satabdi Ghosh, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2019/8875
Record Dates: First submitted 2020-06-25; First posted 2020-07-22 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: MDD
Keywords: Zinc; SSRI; MDD
MeSH Terms: interventions — Selective Serotonin Reuptake Inhibitors; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSRI with placebo (No Intervention): 50 patients who will receive placebo with SSRIs for 8 weeks
- SSRI with zinc sulfate (Active Comparator): 50 patients who will receive SSRIs with zinc sulfate for 8 weeks
  Interventions: Drug: SSRI with Zinc Sulfate

INTERVENTIONS:
Drug: SSRI with Zinc Sulfate — Zinc sulfate (30 mg) once daily for 8 weeks SSRI
  Arms: SSRI with zinc sulfate

SUMMARY:
Title:

Effect of zinc supplementation on depression in SSRIs-treated MDD patients.

Purpose: Depression is the single largest contributor to global disability as has been ranked by WHO (2015), in humans including both male and female.Studies have suggested that conventional presently available anti-depressive medicines are effective for one third to one-half (19-34%) of the patients suffering from depression, leaving the rest of patients to suffer from recurrence or incomplete cure. Researchers throughout the world are involved to obtain new pharmacotherapy for the treatment of MDD. Zinc is an important micronutrient of the human body which is implicated as an essential component in various systemic wellbeing including the central nervous system.

Methods: The study would be randomized, double-blind, placebo-controlled prospective interventional trial and it would be conducted in the Department of Pharmacology and in collaboration with the Department of Psychiatry, BSMMU, from date of approval by the IRB to August 2020. A total of 100 patients suffering from mild to moderate major depression will be selected following to inclusion and exclusion criteria and serum Zinc levels will be assessed. The diagnosis of patients suffering from MDD and the selection of drugs and dosage would be performed by a senior professor of the Psychiatry department. After completing the necessary formalities including the informed consent of the patients, the patient would undergo a selected questionnaire (DASS-21) to assess his/her degree of severity of the disease. The patients would be randomly allocated into two groups: group A (control group) and B (intervention group). Group A would consist of 50 patients who will receive a placebo with SSRIs for 8 weeks. Group B would consist of 50 patients who will receive SSRIs plus Zinc sulfate (30mg/day) orally for 8 weeks, after which at follow up, the severity of depression will be assessed. The blood sample will be collected to measure serum zinc level at baseline and again after 8 weeks of therapeutic intervention.

Ethical consideration

The study will follow the principles of the Declaration of Helsinki and of the World Medical Assembly. Patients will be informed about the study in easy language and then informed consent will be taken. The study has no potential risk to the patients. Confidentiality will be strictly maintained.

DETAILED DESCRIPTION:
Depression (MDD) is a major global health problem. The number of people suffering from major depressive disorder was reported as around 300 million (about 4.4% of the world's population) in 2015. The total number is assumed to increase to 18.4% from 2005 to 2015. Depression is more common in females compared to males (female: male = 5.1:3.6). Years lived with a disability are about 50 million people due to major depressive disorder and this disease has been claimed to be a major cause of morbidity, mortality, and also suicidal death. In Bangladesh, the prevalence of depressive disorder is about 4.1% and the percentage of total years lived with a disability (DALY) is about 7.1%. Within this number, some people suffer additionally from anxiety disorders and some suffer from both anxiety disorder and MDD. However, MDD has been assumed to occupy the place of the second cause of disability by 2020, and MDD, therefore, demands attention and alerts in clinical psychiatry. Depression impairs quality of life at the level of personal, familial, and social aspects and in the severe form, may lead to thoughts of committing suicide. Suicidal death (about 8,00000 per year) have been reported throughout the world in recent reports and are increasing gradually. Conventional antidepressants are the medicines used to treat MDD. Increasing 5HT concentrations at the synapses of the amygdala, frontal cortex, or the limbic region by SSRI or TCA or other drugs administration remains the primary object of therapy. About 19-34% of MDD patients show a reasonable level of response to the SSRIs while about 15-50% of patients show dissatisfactory response or recurrence. This fact is a subject of concern and invite pharmacological intervention either in the form of adjunct drugs or new drug discoveries. Recent researches have revealed that a significant role of zinc in MDD patients due to its antidepressant effects. Some studies reported that there is no effect of zinc supplementation on depression in MDD patients. Because of the conflicted reports, this study has been designed to evaluate the effect of zinc supplementation on depression in MDD patients treated with SSRI. Results of this study may be helpful to advocate the regular use of zinc supplementation as an adjunct to SSRI therapy in MDD. The study would be randomized, double-blind, placebo-controlled prospective interventional trial and it would be conducted in the Department of Pharmacology and in collaboration with the Department of Psychiatry, BSMMU, from the date of approval by the IRB to August 2020. A total of 100 patients suffering from mild to moderate major depression will be selected following to inclusion and exclusion criteria and serum Zinc levels will be assessed. The diagnosis of patients suffering from MDD and the selection of drugs and dosage would be performed by a senior professor of the Psychiatry department. After completing the necessary formalities including the informed consent of the patients, the patient would undergo a selected questionnaire (DASS-21) to assess his/her degree of severity of the disease. The patients would be randomly allocated into two groups: group A (control group) and B (intervention group). Group A would consist of 50 patients who will receive a placebo with SSRIs for 8 weeks. Group B would consist of 50 patients who will receive SSRIs plus Zinc sulfate (30mg/day) orally for 8 weeks, after which at follow up, the severity of depression will be assessed. The blood sample will be collected to measure serum zinc level at baseline and again after 8 weeks of therapeutic intervention. The regularity of medicine intake will be ensured over the telephone, counting the tablets, and from the patient's compliance sheet. The study entails almost no potential risk to the patients which will be explained to the patients together with the fact that he/she would be free to leave the study at any time and that he/she would receive free of cost treatment in case of any adverse reactions. Statistical analysis will be obtained by SPSS (Statistical Package for Social Science). Results will be presented in tables and graphical figures as applicable. Calculated 'p' value may suggest the level of significance (significant at p ≤ 0.050). The study will follow the principles of the Declaration of Helsinki and of the World Medical Assembly. Patients will be informed about the study in easy language and then informed consent will be taken. The study has no potential risk to the patients. Confidentiality will be strictly maintained.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with major depressive disorder diagnosed from the Psychiatry department of BSMMU according to the diagnostic protocol which fulfills DSM-4 criteria and SCID 1 Bangla version.
* Patients treated with only SSRIs.
* Mild to moderate MDD patients.
* Age: 18-55 years.
* Sex: Both male and female.

Exclusion criteria:

* Age < 18 years and > 55 years.
* Patients receiving other antidepressants and dietary supplements in the last two months.
* Patients with other psychiatric disorders (such as anxiety disorder, schizophrenia, bipolar disorder, alcoholism).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
To measure the serum zinc level in SSRI-treated MDD patients pre and post supplementation of zinc. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Satabdi Ghosh, MBBS, Principal Investigator — BSMMU(Recruiting), Dhaka, Bangladesh, 1000
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No